CLINICAL TRIAL: NCT04141410
Title: Levosimendan and Global Longitudinal Strain Assessment in Cardiogenic Shock Sepsis (GLASSES 1): a Study Protocol for an Observational Study
Brief Title: Global Longitudinal Strain Assessment in Cardiogenic Shock During Sepsis
Acronym: GLASSES-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda USL Toscana Centro (Other)
Responsible Party: Principal Investigator, Iacopo Cappellini, Principal Investigator, Azienda USL Toscana Centro
Other Study IDs: 13875 17/18 PO
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Sepsis; Septic Shock; Cardiogenic Shock
Keywords: Sepsis; Septic Shock; Cardiogenic Shock; Speckle Tracking Echocardiography; Levosimendan
MeSH Terms: conditions — Sepsis; Shock, Septic; Shock, Cardiogenic | interventions — Simendan; Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Levosimendan — Use of Levosimendan in cardiogenic shock during sepsis
Device: Echocardiography — Use of global longitudinal strain in cardiogenic shock during sepsis

SUMMARY:
Cardiogenic shock is a condition of low cardiac output that represents the end of a progressive deterioration of cardiac function. The main cause is ischemic heart disease but there are several causes of non-ischemic nature including sepsis.

Sepsis is characterized by a picture of organ dysfunction caused by an altered response of the body to an infection. Its most serious form is septic shock, defined as a picture of sepsis in which the underlying abnormalities in the cardiovascular system and cellular metabolism are such as to increase mortality. An organ failure correlates directly with the function of others and this interdependence is especially evident when a cardiovascular failure is established. 3 Cardiac dysfunction in sepsis can be defined as that of a syndrome characterized by low cardiac output not related to myocardial ischemia.

The use of levosimendan in cardiogenic shock during sepsis was first described in a 2005 case report. Since then there have been small studies and other case reports that have shown improvements in right and left ventricular contractility, ventricular coupling, cardiopulmonary performance, global oxygen transport, renal and splanchnic perfusion when compared to dobutamine and placebo. Other beneficial effects of this drug have emerged, including an anti-inflammatory, antioxidant and antiapoptotic action with a possible protection from ischemia-reperfusion damage.

The present study aims to evaluate the correct use of levosimendan, after the occurrence of cardiogenic shock on a low cardiac index has been ascertained, with the aim of weaning from inotropic drugs in infusion.

DETAILED DESCRIPTION:
The present is an observational single centre no profit study. The duration is expected to be 12 months from September 2019.

The study will be conducted by enrolling patients aged 18 to 80 years in intensive care with diagnosis of septic shock according to the Third National Consensus Definitions for Sepsis and Septic Shock2, with the need for infusion of vasoactive drugs to maintain a PAM > 65 mmHg. The following will be subjected to echocardiographic examination with Sparq ultrasound machine (Philips Healthcare, Best, the Netherlands) and 3.6 MHz cardiology probe through which will be acquired the apical projections 2, 3 and 4 chambers necessary to calculate the global longitudinal strain (GLS) through AutoSTRAIN© (TOMTEC Imaging Systems GmbH, Unterschleissheim, Germany).

During the echocardiographic examination, the Ea/Ees ratio (ventricle-arterial coupling) will also be calculated using the method modified on a single beat of Chen (t0) 18 using the IElastance® application. Patients will be monitored with the PiCCO® system (Pulse index Continuous Cardiac Output, Pulsion Medical systems, Munich, Germany) which measures the cardiac index (CI) and the Stroke Volume Index (SVI). Those with Ea//Ees > 1, cardiac index values < 2.5 L/min/m2 and/or Stroke Volume Index < 30 mL/beat/m2 will be considered eligible to enroll in the study. In these patients, dobutamine infusion will be started from 5 mcg/kg/min following the bundles of the Surviving Sepsis Campaign at dosages that allow to obtain an CI >2.5 L/min/m2 and/or Stroke Volume Index >30 mL/beat/m2. With 24 hours to go before the dobutamine infusion starts, CI and SVI will be recalculated using PiCCO®, GLS and ventricle-arterial coupling index by ultrasound investigation and then levosimendan infusion will begin for 24 hours starting with an infusion of 0.1 mcg/kg/min in order to wean the patient from dobutamine infusion. Once the infusion cycle of the calcium-sensitizing drug has been carried out, if possible, the infusion of dobutamine will be reduced until it stops and CI, SVI, GLS and Ea/Ees will also be re-evaluated. The same echocardiographic evaluations and hemodynamic calculations using PiCCO® will be performed 72 and 96 hours after the start of the dobutamine infusion. All patients enrolled will be followed up by a Medical Outcomes Survey Short-Form 36 (SF-36) questionnaire 28 days and 90 days after discharge from intensive care.

It should be noted that all the procedures described (including echocardiographic monitoring) comply in quantity and frequency with the normal practice of care and management of patients admitted to intensive care with diagnosis of cardiogenic shock during sepsis in Azienda USL Toscana Centro.

In addition, the parameters measured during the echocardiographic examination are derived from the reprocessing of the images collected during the examination and therefore simply represent an in-depth examination for diagnostic purposes performed according to current practice at the Centre.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Age between 18 and 80 years old
* Diagnosis di Sepsis following criteria of Third National Consensus Definitions for Sepsis and Septic Shock 2
* Diagnosis of Cardiogenic Shock with Heart Index < 2.5 L/min/m2 calculated by PiCCO thermodilution method and/or Diagnosis of Stroke Cardiogenic Shock Volume Index < 30 mL/beat/m2 calculated by PiCCO thermodilution method
* Patients applying for treatment with dobutamine and levosimendan according to the procedure laid down in current clinical practice at the Centre
* Ventricle coupling Arterial Ea/Ees > 1 via IElastance application

Exclusion Criteria:

* Age < 18 years and > 80 years
* Pre-existing diagnosis of heart failure at a reduced or preserved ejection fraction
* History of valvular heart disease or valve replacement and/or PM implant
* Severe pulmonary hypertension and chronic pulmonary heart
* Poor acoustic windows for echocardiography
* History of hypersensitivity or allergy to levosimendan

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be those admitted to the intensive care units of the hospital Santo Stefano in Prato with diagnosis of cardiogenic shock during sepsis and who will present the following criteria for inclusion.
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2019-10-21 (Actual); Primary Completion 2020-10-21 (Estimated); Study Completion 2021-01-21 (Estimated)

PRIMARY OUTCOMES:
Global Longitudinal Strain ≥ 15% | up to 1 week
  Recovery of normal values of GLS ≥ 15% after infusion of dobutamine and levosimendan

SECONDARY OUTCOMES:
Mortality | 1 year
  Mortality reduction 30% based on studies where GLS >-15% had half the mortality in those who had a value < 15%.

CONTACTS AND LOCATIONS:
Overall Officials: Iacopo Cappellini, MD, Principal Investigator — Azienda USL Toscana Centro
Locations (1):
- Ospedale Santo Stefano, Prato, FI, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available for 1 year from October 2019

REFERENCES:
- [Derived] Cappellini I, Melai A, Zamidei L, Parise M, Cipani S, Consales G. Levosimendan and Global Longitudinal Strain Assessment in Sepsis (GLASSES 1): a study protocol for an observational study. BMJ Open. 2020 Sep 25;10(9):e037188. doi: 10.1136/bmjopen-2020-037188. PMID 32978191